CLINICAL TRIAL: NCT05350904
Title: Does Hybrid Telehealth Physical Therapy for Children With Moderate to Severe Disability Improve Function in the Home Environment Better Than In-person Services Alone?--A Mixed Methods Study
Brief Title: Hybrid Telehealth in Pediatric Physical Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jamie Hall, Assistant Teaching Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2090371
Record Dates: First submitted 2022-04-05; First posted 2022-04-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Pediatric Disorder; Disability, Developmental
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: The control group will receive usual physical therapy care. The experimental group will receive a hybrid of in-person and telehealth services to address in-home functional skills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hybrid of telehealth and in-person physical therapy services — The experimental group will receive a hybrid of telehealth and in-person physical therapy services to address an in-home functional skill in children with moderate to severe disability.

SUMMARY:
The purposes of this study are to compare the impact of a hybrid of telehealth and in-person physical therapy services to in-person services alone on the in-home functional skills of children with moderate to severe disability. This is a mixed methods study.

DETAILED DESCRIPTION:
The purposes of this study are to compare the impact of a hybrid of telehealth and in-person physical therapy services to in-person services alone on the in-home functional skills of children with moderate to severe disability. Research questions include:

Is a hybrid of telehealth and in-person physical therapy service better than in-person services alone for improving in-home functional skills in children with moderate to severe disability?

Is there a difference in the satisfaction of caregivers and children with physical therapy services which consist of a hybrid of telehealth and in-person physical therapy services compared to in-person services alone?

What is the experience of children and caregivers who receive a hybrid of telehealth and in-person physical therapy services during an episode of care?

ELIGIBILITY:
Inclusion Criteria:

* Children 2-17 years old with moderate to significant disability.
* Families have access to minimum technology necessary to participate in a telehealth visit. ---The child's insurance covers telehealth visits.

Exclusion Criteria:

-Caregiver does not speak English

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure | after physical therapy episode of care an average of 12 weeks
  evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living
Measures of Processes of Care (MPOC) | after physical therapy episode of care, an average of 12 weeks
  Survey tool which assesses parents' perceptions of the care they and their children receive from children's rehabilitation treatment centers. Designed to assess the family-centered behaviours of healthcare providers
Change in Pediatric Evaluation of Disability Inventory | after physical therapy episode of care, an average of 12 weeks
  Assess key functional capabilities and performance in children whose functional abilities are lower than those of seven-year-olds without disabilities
Semi-structured interviews with caregivers and children in experimental group | after physical therapy episode of care, an average of 12 weeks
  Will follow an interview guide designed to capture the experiences of caregivers and children with telehealth

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No